CLINICAL TRIAL: NCT04969354
Title: Clinical Study of CAIX-targeted CAR-T Cells in the Treatment of Advanced Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Collaborators: Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2021-KL092-02
Record Dates: First submitted 2021-07-04; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Immunotherapy
Keywords: Carbonic anhydrase; advanced renal cell carcinoma; CAR-T; Chimeric antigen receptor; T cell; CAIX
MeSH Terms: interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cell immunotherapy (Experimental): The registered patients will received CAR-T cell immunotherapy for the new specific chimeric antigen receptor of CAIX antigen by infusion.
  Interventions: Biological: CAR-T cell immunotherapy

INTERVENTIONS:
Biological: CAR-T cell immunotherapy — This CAR-T cell immunotherapy with a novel specific Chimeric antigen receptor aiming at CAIX antigen.

SUMMARY:
This is an experimental study to evaluate the safety and efficacy of CAR T cells targeting CAIX in the treatment of advanced renal cancer.

DETAILED DESCRIPTION:
We designed a clinical study and divided the trial into two phases.

Phase 1 (climbing test) : 12 patients were randomly divided into 4 groups (n=3). 12 patients were treated with cyclophosphamide at the dose of 60mg/kg/d 8-7 days before CAR-T cell infusion, and fludalabine at the dose of 25mg/m^2/d 6-2 days before CAR-T cell infusion. 5 mg anti-human CAIX monoclonal antibody (G250) was injected into the hepatic artery of each patient by an interventional catheter on the day before CAR-T cells infusion. On Day 0, CAR T cells were injected into patients in group 1, 2, 3 or 4 at the dose of 1x10^7/ person, 1*10^8/ person, 1*10^9/ person or 1*10^10/ person, respectively. The infusion time is about 15-30min. On day 0-14, IL-2 (75000IU/kg) was injected subcutaneously once a day. From day 15-28, IL-2 (75000IU/kg) was subcutaneously injected into the patients three times a week. The purpose of this study is to assess subjects' MTD (maximum tolerated dose) against CAR T cells.

Phase 2: After determining the appropriate therapeutic dose for patients with renal cell carcinoma, 8 patients received the same pre-treatment of chemotherapy and G250 antibody. Then, the appropriate therapeutic dose of CAR T cells according to the results of phase 1 was infused on Day 0. On day 0-14,IL-2 (75000IU/kg) was given subcutaneously once a day. On day 15-28, IL-2 (75000IU/kg) was given subcutaneously three times a week.

Peripheral blood was collected every 4 weeks to evaluate proliferation and survival of CAR-T cells. After 6 months of close follow-up, subjects will undergo a medical history evaluation, physical examination, and blood tests quarterly for 2 years. After this assessment, subjects will be enrolled in an annual telephone follow-up and questionnaire study for up to five years to evaluate treatment for long-term health problems, such as recurrence of malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged from 18 to 70 years old;
2. The patient's ECOG score is ≤ 2;
3. Patients with advanced or metastatic renal cell carcinoma:

(1) have received first-line and second-line targeted therapy in the past; (2) Previous immunization with PD-1/L1 and ≤2 regimens; (3) Unable to tolerate targeted therapy or immunotherapy. 4.There are measurable or evaluable lesions; 5.The main tissues and organs of patients function well:

1. liver function: ALT/AST< 3 times the upper limit of normal value (ULN);
2. Renal function: creatinine < 220 μmol/L;
3. Lung function: indoor oxygen saturation ≥ 95%;
4. Cardiac function: Left ventricular ejection fraction (LVEF)≥40% 6.Patients or their legal guardians voluntarily participate and sign informed consent.

Exclusion Criteria:

1. Infectious diseases (such as HIV, active hepatitis B or C infection, active tuberculosis, etc.);
2. Feasibility assessment and screening showed that the transfection of targeted lymphocytes was less than 10% or the amplification was insufficient (< 5 times) under the co-stimulation of CD3/CD28.
3. The vital signs are abnormal, and those who cannot cooperate with the examination;
4. Those who have mental or psychological diseases can not cooperate with treatment and efficacy evaluation;
5. Highly allergic constitution or severe allergic history, especially those who are allergic to IL-2;
6. Subjects with systemic infection or severe local infection who need anti-infection treatment;
7. Complicated with dysfunction of heart, lung, brain, liver, kidney and other important organs;
8. Patients with other tumors;
9. Doctors believe that there are other reasons that can not be included in the treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation:Incidence and severity of adverse events | First 1 month after CAR-T cells infusion
  To evaluate the incidence and severity of possible adverse events within one month after targeted CAIX CAR-T infusion, including cytokine release syndrome and on-target toxicity.
Effectiveness evaluation | 3 months after CAR-T cells infusion
  In order to observe the efficacy of CAR-T cells after infusion, total remission rate (ORR), complete remission (CR), partial remission (PR), disease stability (SD) or progression (PD) will be used for evaluation.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 24 months after CAR-T cells infusion
  Progression-free survival (PFS) time
Overall survival (OS) | 24 months after CAR-T cells infusion
  Overall survival (OS) time

CONTACTS AND LOCATIONS:
Overall Officials: Junnian Zheng, M.D/Ph.D, Study Director — The Affiliated Hospital of Xuzhou Medical University; Hailong Li, M.D/Ph.D, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University; Qing Zhang, Ph.D, Principal Investigator — Xuzhou Medical University
Locations (1):
- Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Linehan WM, Ricketts CJ. Kidney cancer in 2016: RCC - advances in targeted therapeutics and genomics. Nat Rev Urol. 2017 Feb;14(2):76-78. doi: 10.1038/nrurol.2016.260. Epub 2016 Dec 29. No abstract available. PMID 28031562
- [Result] Zhang Q, Li H, Yang J, Li L, Zhang B, Li J, Zheng J. Strategies to improve the clinical performance of chimeric antigen receptor-modified T cells for cancer. Curr Gene Ther. 2013 Feb;13(1):65-70. doi: 10.2174/156652313804806570. PMID 23256743
- [Result] Sadelain M, Riviere I, Riddell S. Therapeutic T cell engineering. Nature. 2017 May 24;545(7655):423-431. doi: 10.1038/nature22395. PMID 28541315
- [Result] Xu J, Tian K, Zhang H, Li L, Liu H, Liu J, Zhang Q, Zheng J. Chimeric antigen receptor-T cell therapy for solid tumors require new clinical regimens. Expert Rev Anticancer Ther. 2017 Dec;17(12):1099-1106. doi: 10.1080/14737140.2017.1395285. Epub 2017 Oct 26. PMID 29048935
- [Result] Weinkove R, George P, Dasyam N, McLellan AD. Selecting costimulatory domains for chimeric antigen receptors: functional and clinical considerations. Clin Transl Immunology. 2019 May 11;8(5):e1049. doi: 10.1002/cti2.1049. eCollection 2019. PMID 31110702
- [Result] Brentjens RJ, Davila ML, Riviere I, Park J, Wang X, Cowell LG, Bartido S, Stefanski J, Taylor C, Olszewska M, Borquez-Ojeda O, Qu J, Wasielewska T, He Q, Bernal Y, Rijo IV, Hedvat C, Kobos R, Curran K, Steinherz P, Jurcic J, Rosenblat T, Maslak P, Frattini M, Sadelain M. CD19-targeted T cells rapidly induce molecular remissions in adults with chemotherapy-refractory acute lymphoblastic leukemia. Sci Transl Med. 2013 Mar 20;5(177):177ra38. doi: 10.1126/scitranslmed.3005930. PMID 23515080
- [Result] Song C, Sadashivaiah K, Furusawa A, Davila E, Tamada K, Banerjee A. Eomesodermin is required for antitumor immunity mediated by 4-1BB-agonist immunotherapy. Oncoimmunology. 2014 Jan 1;3(1):e27680. doi: 10.4161/onci.27680. Epub 2014 Feb 27. PMID 24790793
- [Result] Maude SL, Frey N, Shaw PA, Aplenc R, Barrett DM, Bunin NJ, Chew A, Gonzalez VE, Zheng Z, Lacey SF, Mahnke YD, Melenhorst JJ, Rheingold SR, Shen A, Teachey DT, Levine BL, June CH, Porter DL, Grupp SA. Chimeric antigen receptor T cells for sustained remissions in leukemia. N Engl J Med. 2014 Oct 16;371(16):1507-17. doi: 10.1056/NEJMoa1407222. PMID 25317870
- [Result] Kawalekar OU, O' Connor RS, Fraietta JA, Guo L, McGettigan SE, Posey AD Jr, Patel PR, Guedan S, Scholler J, Keith B, Snyder NW, Blair IA, Milone MC, June CH. Distinct Signaling of Coreceptors Regulates Specific Metabolism Pathways and Impacts Memory Development in CAR T Cells. Immunity. 2016 Mar 15;44(3):712. doi: 10.1016/j.immuni.2016.02.023. Epub 2016 Mar 15. No abstract available. PMID 28843072
- [Result] Long AH, Haso WM, Shern JF, Wanhainen KM, Murgai M, Ingaramo M, Smith JP, Walker AJ, Kohler ME, Venkateshwara VR, Kaplan RN, Patterson GH, Fry TJ, Orentas RJ, Mackall CL. 4-1BB costimulation ameliorates T cell exhaustion induced by tonic signaling of chimeric antigen receptors. Nat Med. 2015 Jun;21(6):581-90. doi: 10.1038/nm.3838. Epub 2015 May 4. PMID 25939063
- [Result] Lamers CH, Sleijfer S, van Steenbergen S, van Elzakker P, van Krimpen B, Groot C, Vulto A, den Bakker M, Oosterwijk E, Debets R, Gratama JW. Treatment of metastatic renal cell carcinoma with CAIX CAR-engineered T cells: clinical evaluation and management of on-target toxicity. Mol Ther. 2013 Apr;21(4):904-12. doi: 10.1038/mt.2013.17. Epub 2013 Feb 19. PMID 23423337
- [Result] Lamers CH, Willemsen R, van Elzakker P, van Steenbergen-Langeveld S, Broertjes M, Oosterwijk-Wakka J, Oosterwijk E, Sleijfer S, Debets R, Gratama JW. Immune responses to transgene and retroviral vector in patients treated with ex vivo-engineered T cells. Blood. 2011 Jan 6;117(1):72-82. doi: 10.1182/blood-2010-07-294520. Epub 2010 Oct 1. PMID 20889925